CLINICAL TRIAL: NCT05690685
Title: Post-market Surveillance Study to Confirm the Safety and Performance of Silver I Alginate Non-Woven Dressing (Hydro-Alginate) in Chronic and Acute Wounds
Brief Title: PMS Study of Silver I Alginate Non-Woven Dressing (Hydro-Alginate)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Silver I Alginate NonWoven 001
Record Dates: First submitted 2022-12-21; First posted 2023-01-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Silver I Alginate Non-Woven Dressing (Hydro-Alginate) (Experimental): Subjects will undergo treatment of their chronic or acute wound (Pressure ulcer, and Donor sites) as indicated in the instructions for use with Silver I Non-Woven Dressing
  Interventions: Device: Silver I Alginate Non-Woven Dressing (Hydro-Alginate)

INTERVENTIONS:
Device: Silver I Alginate Non-Woven Dressing (Hydro-Alginate) — Assigned interventions Subjects will undergo treatment of their chronic and acute wounds as indicated in instructions for use with Silver I Non-Woven dressings.
  Subjects will be evaluated as follows:
  Full Patient and wound assessment, Informed consent. Wound Assessment, application of dressings, (At each scheduled dressing change.) Wound Assessment, removal of dressings, (At each scheduled dressing change.) The patients will be evaluated at each dressing change up-to six-week follow-up period.
  Other Names: Silvercel (brand name)

SUMMARY:
Post market surveillance study to confirm the ongoing safety and performance of Silver I Alginate Non-Woven Dressing (Hydro-Alginate) in chronic and acute wounds.

DETAILED DESCRIPTION:
Design: The design of the study is an open-label, multicentre, single arm clinical trial in subjects with moderate to heavily exuding chronic and acute wounds consisting of Pressure ulcers and Donor sites.

The rationale for the chosen study design and objectives is based on the requirement for further confirmation of the clinical effectiveness and safety of the dressing in routine clinical use, in terms of management of wound, management of bioburden, maintaining a moist wound environment, and exudate management.

This post market study has been designed to be an in-market clinical evaluation. Using the assessment scale of "satisfactory" or "not satisfactory" will indicate whether the device is acceptable to the Healthcare Professional and therefore demonstrate the acceptability of the Silver I Alginate Non-Woven dressing (Hydro-Alginate).

It is intended to recruit 25-30 subjects per wound type in support of providing evidence of effectiveness and safety of wound dressings. The prior CE-marking evaluation for this device lacked information pertaining to the use of the device in pressure ulcers or donor site wounds. Therefore, this study will address this gap. This study analysis will be descriptive in nature, for each wound type and will not be based on any stand-alone statistical hypotheses.

The study endpoints have been chosen because they will demonstrate the safety and effectiveness of the dressing in routine clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 18 years or above. (Females must not be pregnant and if of reproductive age should provide a negative pregnancy test at screening).
2. Patients who are able to understand and give informed consent to take part in the study.
3. Have one or more of the following: Pressure ulcer or Donor site wounds that are infected, or are at high risk of infection (in the opinion of the Investigator), that are moderate to heavy levels of exudate.
4. Pressure ulcers that are moderate to high exudate, typically Category 3 and 4.
5. Only one primary wound may be treated per patient for the study.

Exclusion Criteria:

1. Patients who are known to be non-compliant with medical treatment,
2. Patients who are known to be sensitive to any of the device components
3. Subject is pregnant or actively breastfeeding;
4. Subject has a known sensitivity to Silver;
5. Life expectancy of <6 months;
6. Subject has any significant or unstable medical or psychiatric condition that, in the opinion of the Investigator, would interfere with his/her ability to participate in the study;
7. Subject is currently enrolled in another clinical study, or has completed a clinical study less than 30 days prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of Wound progression following 6 weeks (Efficacy) | 6 weeks
  wound progression from baseline to end of follow-up.
  In order to be considered successful in wound progression, at least one of the following must occur in the change from baseline to the end of follow-up:
  * Increase in % of wound granulation tissue
  * Decrease in wound size (volume, area, or depth) or wound closure
  * Decrease in devitalized tissue
  In addition to the following:
  • Reduction or no signs or symptoms of clinical infection.
Subject incidence of any treatment-related adverse events during follow-up period - 6 weeks (Safety) | 6 weeks
  The primary safety analysis will be the calculation of the subject incidence of any treatment-related adverse events between treatment initiation and the end of follow-up for each patient.

SECONDARY OUTCOMES:
Pain assessment | 6 weeks
  Change in patient pain (using Visual Analog Score for pain-VAS Score) from baseline to end of follow-up.
  Min-Max VAS score: 0=no pain to 10=worst pain imaginable. Higher pain VAS score would mean a worse outcome.
Change in wound odour | 6 weeks
  Change in wound odour (using Verbal Numeric Scale- VNS score), from baseline to end of follow-up.
  Min-Max score: 0= no odour to 4= Smell is present but is perceived as extremely offensive.
  A higher odour VNS score would mean a worse outcome.
Ease of use assessment using Likert-type scale | 6 weeks
  Clinician satisfaction with the device (conformability and ease of use) will be assessed using a Likert-type scale.
  Min-Max score: 1=Very easy to 5=Very difficult. A higher score would mean a worse outcome.
Change in wound granulation tissue | 6 weeks
  Change in % of wound granulation tissue.
Percent change in wound size | 6 weeks
  Percent change in wound size (% change in: volume, area or depth).
Percent change in devitalized tissue | 6 weeks
  Percent change in devitalized tissue
Rates of individual components of wound progression (primary efficacy endpoint) | 6 weeks
  Rates of individual components of the primary efficacy endpoint, including:
  * Increase in % of wound granulation tissue
  * Decrease in wound size (volume, area, or depth) or wound closure
  * Decrease in devitalized tissue
  * Reduction or no signs or symptoms of clinical infection.
  For each of these components, the frequency and proportion of successes will be calculated for each wound type.
The number of components of the primary efficacy endpoint experienced by each subject | 6 weeks
  Descriptive statistics of the number of components of the primary efficacy endpoint experienced by each subject, including:
  * Increase in % of wound granulation tissue
  * Decrease in wound size (volume, area, or depth) or would closure
  * Decrease in devitalized tissue
  * Reduction or no signs or symptoms of clinical infection
  For each subject, the number of successful primary efficacy endpoint components will be calculated (range: 0 - 4). Subjects missing data on any of the four primary efficacy endpoint components will be excluded from this secondary endpoint analysis. Descriptive statistics will be provided for the number of successful primary efficacy endpoint components for each wound type, treating the number of components as a continuous variable.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal United Hospital Bath, Bath
  - Queen Victoria Hospital, East Grinstead

IPD SHARING:
Plan to Share IPD: No